CLINICAL TRIAL: NCT06245447
Title: Brain MRI Longitudinal Volumetric Characteristics Associated With Outcomes of CASPR2-Limbic Encephalitis
Acronym: C2-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0106
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Autoimmune Encephalitis Associated With Anti-CAPR2 Antibodies
Keywords: Autoimmune encephalitis, CASPR2 antibodies, MRI
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASPR2- Patients
  Interventions: Other: Retrospective evaluation of specific brain MRI features
- Patients affected by autoimmune encephalitis with antibodies against CASPR2
  Interventions: Other: Retrospective evaluation of specific brain MRI features

INTERVENTIONS:
Other: Retrospective evaluation of specific brain MRI features — * Brain MRI changes in the acute stage, i.e. < 3 months from symptoms onset, including abnormal signal intensity, altered diffusion and/or contrast enhancement in the hippocampus (unilateral/bilateral), abnormal signal intensity in basal ganglia, insula, and/or perisylvian cortex, presence of global brain atrophy, presence of hippocampal atrophy and/or MTS, hippocampal volumetry
  * Brain MRI changes after acute phase resolution (> 6 months after symptoms onset) including abnormal signal intensity in the hippocampus (unilateral/bilateral), presence of global brain atrophy, presence of hippocampal atrophy and/or MTS, hippocampal volumetry

SUMMARY:
Anti-CASPR2 limbic encephalitis (CASPR2-LE) is a rare neurological disorder primarily affecting males over the age of 50. It is mediated by an autoimmune antibody response in the central nervous system (CNS) against the cellular adhesion molecule contactin-associated protein-like 2 (CASPR2). This protein plays an important role in the trafficking of KV1 channels under the myelin sheath in the juxtaparanodal region of myelinated axons. It is mostly present in the neurons of the limbic system, basal ganglia, and other motor related and sensation areas (Qin, Yang, Zhu, Wang, & Shan, 2021). This distribution explains the diverse clinical manifestations of the disease, primarily characterized by cognitive impairment. Other manifestations include cerebellar ataxia, hyperkinetic movement disorders (HMDs), seizures, and neuropathic pain, which all typically develop around 10.4 months after onset. At last visit, memory impairment is seen in 69% of the patients, cerebellar ataxia in 42% of the patients, and functional dependency in 25% of the patients. Even though most patients' symptoms improve with immune-active treatments, up to 69% of them have long-term memory impairments due to damage to hippocampal structures (Benoit et al., 2023). Research has primarily focused on understanding the disease's clinical features, underlying mechanisms, and potential treatment options. On the other hand, it is shown that MRIs performed at baseline show signal changes in the hippocampus in 62-71% of the patients, and these changes are subject to variations in subsequent follow-up scans, that differ widely among patients as mentioned before (Bien et al., 2017). And since the dynamics of hippocampal volume changes and its association with the development of hippocampal atrophy and long-term cognitive impairment are not well studied yet in CASPR2-LE, we primarily aim to examine the longitudinal changes of hippocampal volume in anti-CASPR2 Limbic Encephalitis (CASPR2-LE) patients to examine whether it correlates to the development of anterograde amnesia and hippocampal atrophy on follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite diagnosis of CASPR2-antibody-associated encephalitis
* available MRI records
* Ascertained positivity for CASPR2-antibodies in CSF

Exclusion Criteria:

* Positivity for another antibody against neural or glial antigens
* MRI images not available
* Not enough clinical data to ascertain outcome

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included from the from the database of the French Reference Centre for Paraneoplastic Neurological Syndromes and Autoimmune Encephalitis (Lyon, France)
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Functional independance | 12 months after first treatment
  Defined by a modified Rankin Scale (mRS) score ≤2

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France